CLINICAL TRIAL: NCT01683370
Title: Pediatric FN Definition 2012 Bern The Impact of Lowering Fever Limits on the Rate of Fever in Chemotherapy-induced Neutropenia (FN). A Prospective Single-center Observational Study in Children and Adolescents With Cancer.
Brief Title: Pediatric FN Definition 2012 Bern
Status: Completed | Type: Observational
Sponsor: Dr. Roland Ammann (Other)
Collaborators: Swiss Cancer League (Other)
Responsible Party: Sponsor-Investigator, Dr. Roland Ammann, Associate Professor, Swiss Pediatric Oncology Group
Organization: Swiss Pediatric Oncology Group (Other)
Other Study IDs: PFND2012B; KFS-2933-02-2012 (Other Grant/Funding Number: Krebsforschung Schweiz)
Record Dates: First submitted 2012-08-31; First posted 2012-09-11 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Cancer in Children/Adolescents; Fever in Neutropenia
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1 mL serum, kept refrigerated until the end of study, then analyed as batch for cortisol, then discarded.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Pediatric patients with cancer, receiving standard chemotherapy, and receiving standard supportive therapy in case of fever in neutropenia (FN) (No intervention for study purposes)

SUMMARY:
STUDY AIMS Based on prospectively collected information on ear temperatures, ANC values, emergency calls and consultations for fever, and on hospitalizations for FN in children and adolescents with cancer

* to describe the frequency of episodes of FN, and of other clinically relevant FN-related measures
* to compare these frequencies and measures in reality vs. applying Bernese standard limits for defining fever (ear temperature ≥39.0°C)
* to compare these frequencies and measures applying the Bernese standard limit of ≥39.0°C (LimitStandard) vs. a range of hypothetically lower limits defining fever (LimitLow)
* to determine if it would be useful to perform an interventional study on the question of different fever limits, powered to study both efficacy (frequency of FN) and safety (AE in delayed FN diagnosis)
* to use the platform of this prospective study to explore if the serum level of cortisol is associated with adverse events in FN

HYPOTHESIS In children and adolescents with cancer, hypothetically modifying the definitions of fever from ear temperature 39.0°C to lower limits would

* increase the rate of FN episodes diagnosed during chemotherapy (primary endpoint).
* increase the rate of other clinically important FN-related measures related to chemotherapy exposure time (secondary endpoints 1,2,3) and outcome/treatment-related measures during treatment of FN episodes diagnosed in reality (secondary endpoints 4,5,6).
* not relevantly decrease the proportion of FN with AE (secondary endpoint 7).

ELIGIBILITY:
Inclusion Criteria:

* >1 year and ≤17 years at time of recruitment
* Chemotherapy treatment because of any malignancy for at least 2 months at time of recruitment
* Written informed consent from patients and/or parents for the study

Exclusion Criteria:

* Infants ≤1 year old (reason: differences in standard fever limit and method to measure temperature)
* Denied written informed consent from patients and/or parents for the study

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients diagnosed with cancer requiring chemotherapy, treated at the Division of Pediatric Hematology/Oncology, Department of Pediatric, University of Bern / Inselspital, CH-3010 Bern, Switzerland
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Rate ratio of additional episodes of FN diagnosed (applying LimitLow vs. LimitStandard) | until 2 weeks after last dose of chemotherapy (expected median, 6 months)

SECONDARY OUTCOMES:
Rate of episodes of fever | until 2 weeks after last dose of chemotherapy (expected median, 6 months)
  (Protocol: 1)
Rate of emergency calls for fever | until 2 weeks after last dose of chemotherapy (expected median, 6 months)
  (Protocol: 2a)
Rate ratio of FN diagnosed earlier (applying LimitLow vs. LimitStandard) | until 2 weeks after last dose of chemotherapy (expected median, 6 months)
  (Protocol: 3)
Proportion of FN with blood cultures performed after start of antibiotics (AB) for prolonged fever | until end of AB therapy for FN (estimated median, 4 days)
  (Protocol: 4a)
Proportion of FN with delayed hospital discharge for prolonged fever | until end of AB therapy for FN (estimated median, 4 days)
  (Protocol: 5) (Low risk FN episodes with first-day stepping down will be excluded from this analysis.)
Time point of empirical AB switch for prolonged fever during FN | until end of AB therapy for FN (estimated median, 4 days)
  (Protocol: 6a)
Proportion of FN with any adverse event | until end of AB therapy for FN (estimated median, 4 days)
  (Protocol: 7a)
Serum level of cortisol | at presentation with FN (in reality)
  (Protocol: 8)
Proportion of FN with switch of empirical AB for prolonged fever | until end of AB therapy for FN (estimated median, 4 days)
  (Protocol: 4b)
Proportion of FN with add-on of empirical antifungal therapy for prolonged fever | until end of AB therapy for FN (estimated median, 4 days)
  (Protocol: 4c)
Rate of emergency CBC with consultation for fever | until 2 weeks after last dose of chemotherapy (expected median, 6 months)
  (Protocol: 2b)
Time point of starting empirical antifungal therapy for prolonged fever during FN | until end of AB therapy for FN (estimated median, 4 days)
  (Protocol: 6b)
Proportion of FN with bacteremia | until end of AB therapy for FN (estimated median, 4 days)
  (Protocol: 7b)
Proportion of FN with serious medical complication | until end of AB therapy for FN (estimated median, 4 days)
  (Protocol: 7c)

CONTACTS AND LOCATIONS:
Overall Officials: Roland A Ammann, MD, Study Chair — Pediatric Hematology/Oncology, Department of Pediatrics, University of Bern, Bern, Switzerland
Locations (1):
- Division of Hematology/Oncology, Department of Pediatrics, University of Bern / Inselspital, Bern, Switzerland

REFERENCES:
- [Result] Ammann RA, Teuffel O, Agyeman P, Amport N, Leibundgut K. The influence of different fever definitions on the rate of fever in neutropenia diagnosed in children with cancer. PLoS One. 2015 Feb 11;10(2):e0117528. doi: 10.1371/journal.pone.0117528. eCollection 2015. PMID 25671574
- [Result] Wagner S, Brack EK, Stutz-Grunder E, Agyeman P, Leibundgut K, Teuffel O, Ammann RA. The influence of different fever definitions on diagnostics and treatment after diagnosis of fever in chemotherapy-induced neutropenia in children with cancer. PLoS One. 2018 Feb 20;13(2):e0193227. doi: 10.1371/journal.pone.0193227. eCollection 2018. PMID 29462193
- [Result] Brack E, Wagner S, Stutz-Grunder E, Agyeman PKA, Ammann RA. Temperatures, diagnostics and treatment in pediatric cancer patients with fever in neutropenia, NCT01683370. Sci Data. 2020 May 26;7(1):156. doi: 10.1038/s41597-020-0504-9. PMID 32457478
- [Result] Lavieri L, Koenig C, Teuffel O, Agyeman P, Ammann RA. Temperatures and blood counts in pediatric patients treated with chemotherapy for cancer, NCT01683370. Sci Data. 2019 Jul 3;6(1):108. doi: 10.1038/s41597-019-0112-8. PMID 31270328